CLINICAL TRIAL: NCT02893189
Title: Chimeric Antigen Receptor (CAR)19 Donor Lymphocytes for Relapsed Cluster of Differentiation (CD)19+ Malignancies Following Allogeneic Transplantation (CARD)
Brief Title: CAR19 Donor Lymphocytes for Relapsed CD19+ Malignancies Following Allogeneic Transplantation
Acronym: CARD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL16/0045
Record Dates: First submitted 2016-05-17; First posted 2016-09-08 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: CD19+ Malignancies: Relapse Post-allogeneic Transplant
Keywords: CD19+; allogeneic transplant; relapse
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4G7-CARD T-cells (Experimental): All patient will receive modified CAR19 T-cells.
  Interventions: Genetic: Infusion of modified CAR19 T-cells (4G7-CARD T-cells)

INTERVENTIONS:
Genetic: Infusion of modified CAR19 T-cells (4G7-CARD T-cells) — The original stem cells donor (or if not available the patient) will undergo unstimulated leucapheresis for generation of the Advanced Therapy Interventional Medicinal Product (ATIMP) 4G7-CARD T-cells. Escalating doses of the ATIMP will then be infused to the patient depending on outcome and any experienced side effects.

SUMMARY:
Eligible patients will receive escalating doses of 4G7-CARD T-cells paralleling clinical standard of care with unmanipulated donor lymphocytes. There are 3 intra-patient dose levels planned.

Patients will be followed up regularly during the interventional phase of the study until 12 months post-final 4G7-CARD T-cell infusion. Thereafter patients will be followed up annually for years 2 and 3.

DETAILED DESCRIPTION:
Patients will receive escalating doses of 4G7-CARD T-cells (after pre-conditioning with Fludarabine and Cyclophosphamide), paralleling clinical standard of care with unmanipulated donor lymphocytes. Intra-patient dose escalation will proceed at intervals of not less than 8 weeks, dependent on development of toxicity or evidence of efficacy and confirmation by the Trial Management Group.

Three dose cohorts levels are planned, and dosing will be according to total CD3+ T- cell dose as this correlates with toxicity in the unmanipualated donor lymphocyte setting:

* Dose Level 1: 1x10^6 CD3+ T-cells/kg (starting dose for all patients)
* Dose Level 2: 3x10^6 CD3+ T-cells/kg
* Dose Level 3: 1x10^7 CD3+ T-cells/kg

The inter-patient dosing for the first 3 patients was at least 28 days, following TMG confirmation.

Patients will be followed up regularly during the interventional phase of the study until 12 months post-final 4G7-CARD T-cell infusion. During the long term follow up phase of the study (years 2-3 post-final 4G7-CARD T-cell infusion) patients will be followed-up annually for overall survival, disease status and safety.

All patients will enter long term follow up until 3 years post-final 4G7-CARD T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-70 years
2. Confirmed diagnosis of CD19+ malignancy relapsing following allogeneic transplantation
3. Agreement to have a pregnancy test, use adequate contraception for 12 months post-final 4G7-CARD T-cell infusion
4. Karnofsky performance status >60
5. Written informed consent

Exclusion Criteria:

1. Women who are pregnant or lactating
2. Prior history of ischaemic heart disease, dysrhythmias, abnormal ECG (LBBB), Multi Gated Acquisition Scan (MUGA) left ventricular ejection fraction (LVEF<40%) (if performed)
3. Known involvement of the central nervous system or cerebral vascular accident within prior 3 months
4. Patients receiving corticosteroids at a dose of > 10mg prednisolone per day (or equivalent)
5. Active graft versus host disease requiring immunosuppression
6. Use of rituximab within the last 2 months prior to ATIMP infusion
7. Known allergy to albumin or dimethyl sulfoxide (DMSO)
8. Patients who have experienced significant neurotoxicity following blinatumomab treatment

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of generation of 4G7-CARD T-cells using the ProdigyTM system | Through patient registration and manufacturing period, an average of 18 months from start of trial
  The number of ATIMP successfully manufactured would be assessed for all registered patients
Maximum grade for each toxicity type as assessed by CTCAE v4.03, summarized as proportions. | Up to 3 years post final 4G7-CARD T-cell infusion
  Toxicity evaluation following 4G7-CARD T-cell administration as evaluated by the occurrence of adverse events per studied dose using CTCAE v4.03, defined as >grade 2 events that are causally related to study treatment or procedure or Serious Adverse Reactions that require withdrawal of the patient from the study; development and severity of graft-versus-host-disease (GvHD) following cell infusion will also be evaluated as a potential toxicity, as well as development and severity of cytokine release syndrome / macrophage activation syndromes assessed by 'University of Pennsylvania' criteria

SECONDARY OUTCOMES:
Assessment of engraftment, expansion and persistence of the 4G7-CARD T-cells as determined by quantitative polymerase chain reaction (qPCR) or flow cytometry | Sampling occurs at days 0, 4, 6, 11, 18, plus months 1, 2, 3, 6, 9 and 1 year post final 4G7-CARD T-cell infusion
  Data for engraftment and expansion would be summarised by mean, median or interquartile ranges and a Kaplan Meier plot for persistence
Assessing the depletion of B cell compartment, as determined by flow cytometry | Sampling occurs at days 0, 4, 6, 11, 18, plus months 1, 2, 3, 6, 9 and 1 year post final 4G7-CARD T-cell infusion
  Data would be summarised using means (medians) and as the percentage reduction from baseline
Assessing the timing and magnitude of cytokine release, evaluated using Cytokine bead arrays | Sampling occurs at days 0, 4, 6, 11, 18, plus 1 month post final 4G7-CARD T-cell infusion
  Data on timing (kinetic of change) and magnitude of cytokine levels can be summarised using means (medians) and plots for each patients

CONTACTS AND LOCATIONS:
Overall Officials: Karl Peggs, Principal Investigator — University College London Hospital
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roddie C, Dias J, O'Reilly MA, Abbasian M, Cadinanos-Garai A, Vispute K, Bosshard-Carter L, Mitsikakou M, Charalambous E, Mehra V, Roddy H, Cheung GW, Hartley JA, Mahmoud N, Ensell L, Patel Y, Marzolini MAV, Farzaneh F, Nickolay L, Himoudi N, Syed F, Popova B, Galani S, Day A, Lowdell MW, Peggs KS. Matched donor allogeneic CAR-T for adult B-ALL: toxicity, efficacy, repeat dosing, and the importance of lymphodepletion. Blood. 2025 Oct 2;146(14):1664-1676. doi: 10.1182/blood.2025028790. PMID 40643148
- [Derived] O'Reilly M, Roddie C, Marzolini MAV, Rodriguez-Justo M, Pomplun S, Pule M, Peggs KS. Trafficking of CAR T cells to sites of subclinical leukaemia cutis. Lancet Oncol. 2020 Mar;21(3):e179. doi: 10.1016/S1470-2045(19)30861-7. No abstract available. PMID 32135121